CLINICAL TRIAL: NCT07046832
Title: Clinical Evaluation of an Intra-procedural 3D Needle Guidance Platform for Soft Tissue Tumors or Organs Requiring Percutaneous Biopsy as an Adjunct to Standard Image Guidance
Brief Title: Clinical Evaluation of an Augmented Reality Intraprocedural Needle Guidance Platform for Soft Tissue Biopsy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: MediView XR, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 24-06-433
Record Dates: First submitted 2025-06-13; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Oncology; Interventional Radiology; Liver Carcinoma; Renal Carcinoma; Biopsy
Keywords: Percutaneous Interventions; Needle Guidance; Augmented Reality; Medical Device; XR90; Minimally Invasive
MeSH Terms: conditions — Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Renal Cell

STUDY DESIGN:
Intervention Model Description: Multicenter prospective randomized control trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Arm A, XR90 (Experimental Group) (Experimental): Participants randomly assigned to this arm will undergo percutaneous biopsy procedures using the assistance of XR90 guidance system in adjunct to standard of care guidance.
  Interventions: Device: Augmented Reality Guided Biopsy
- Arm B (Standard of Care Group) (Active Comparator): Participants randomly assigned to this arm will undergo percutaneous biopsy with standard of care CT and ultrasound needle guidance only.
  Interventions: Device: Ultrasound Guided Biopsy

INTERVENTIONS:
Device: Augmented Reality Guided Biopsy — Augmented Reality system in adjunct to standard of care guidance for needle guidance during a percutaneous biopsy
  Arms: Arm A, XR90 (Experimental Group)
Device: Ultrasound Guided Biopsy — Ultrasound guided biopsy as a part of standard of care.
  Arms: Arm B (Standard of Care Group)

SUMMARY:
This clinical feasibility evaluation is intended to further characterize and quantify the potential benefits of the FDA-cleared XR90 Augmented Reality (AR )imaging and guidance platform utilization in percutaneous soft tissue biopsy. This study will seek to build on the findings of safety, procedural benefits, and overall clinical feasibility shown in previous bench, cadaveric, and single-site clinical evaluations.

DETAILED DESCRIPTION:
This clinical evaluation is needed to further characterize and quantify the potential benefits of percutaneous biopsy, assisted with the XR90 3D surgical imaging system. This continued innovative implementation of the platform as a medical device to assist in percutaneous targeted biopsy of soft tissue tumors will allow for further assessment of device functionality, operator acceptability, and additional data collection to help quantify the potential benefits of this platform. Potential benefits to the patient, to be formally proven in future studies: decreased procedure time, decreased of complications (e.g., critical structure avoidance), and ultimately, improved patient outcomes. To date, few studies have evaluated the performance of the XR90 guidance system in a clinical setting. Comparing percutaneous needle placement for biopsies of a soft tissue target with the assistance of XR90 compared to under only standard-of-care guidance will allow for the evaluation of procedure success rate, overall procedure time, and complications. This multicenter prospective randomized control trial is designed to compare the efficacy and utility of the XR90 guidance platform used adjunct to standard of care guidance to standard of care guidance (2D) only for percutaneous needle-based procedures.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Willing and able to give informed consent prior to enrollment
* Subjects in need of a diagnostic soft-tissue tumor biopsy which is the primary target for needle placement as a part of their standard of care.
* Subjects who have met all criteria to undergo percutaneous biopsy with ultrasound.
* Subjects with soft-tissue lesions ≥1 cm or ≤8 cm in depth
* BMI of ≤40

Exclusion Criteria:

* Children under the age of 18.
* Currently pregnant at the time of the procedure
* Not willing or able to give informed consent.
* Subjects with pacemakers or AICDs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Time of Tumor Localization | Intraprocedural-from the start of the procedure until the end of the study procedure, 1 day.
  The time from initiation of localization of imaging (defined by when the ultrasound probe is put into operator's hand) until operator has planned a trajectory and point of entry (by placing a finger or trocar on the skin entry site and verbalizing completion of localization) will be measured and recorded. Time is recorded in minutes and will be completed during the procedure.
Time From Skin to Target | Intraprocedural, from the start of the procedure until the end of the study procedure, 1 day.
  The elapsed time from when the proceduralist inserts their trocar or biopsy needle through the skin (excluding skin knicks) and when the provider verbalizes they have reached their intended target in order to collect a biopsy under ultrasound guidance. Time will be recorded in minutes beginning and ending during the study procedure.

SECONDARY OUTCOMES:
Technical Success | Duration of the study procedure
  The completion of the biopsy procedure. Procedures will be determined to be complete once the provider has verified (via ultrasound or CT) the trocar has reached the intended target, as if the proceduralist were to ablate or biopsy
Needle Attempts | Duration of the study procedure
  An attempt will be counted at the beginning of targeting and each time an operator removes their needle from the skin and restarts localization.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - MedStar Georgetown Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hosptial Center, Washington D.C., District of Columbia
  - NewYork-Presbyterian Weill Cornell Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No
The trial evaluates a novel augmented reality needle guidance platform that includes investigational software features and procedural performance data. These elements are considered proprietary and form part of an active product development that may be incorporated as part of a broader regulatory strategy.
  In addition, the study's small sample size and highly structured procedural metrics - including EM tracking outputs, intraoperative timing, and device-specific workflow parameters - increase the risk of participant re-identification, even without direct identifiers or imaging.
  To protect intellectual property and ensure compliance with HIPAA, GDPR, and FDA confidentiality provisions (21 CFR § 812.38; 21 CFR § 20.61), individual participant data (IPD) will not be shared. Summary-level data and aggregate results will be made available through peer-reviewed publications and posted on ClinicalTrials.gov

REFERENCES:
- [Background] Al-Nimer S, Hanlon A, Cho K, Kalra-Lall A, Weunski C, Yanof J, West K, Martin C 3rd. 3D Holographic Guidance and Navigation for Percutaneous Ablation of Solid Tumor. J Vasc Interv Radiol. 2020 Mar;31(3):526-528. doi: 10.1016/j.jvir.2019.09.027. Epub 2020 Jan 31. No abstract available. PMID 32008844
- [Background] Gadodia G, Yanof J, Hanlon A, Bustos S, Weunski C, West K, Martin C 3rd. Early Clinical Feasibility Evaluation of an Augmented Reality Platform for Guidance and Navigation during Percutaneous Tumor Ablation. J Vasc Interv Radiol. 2022 Mar;33(3):333-338. doi: 10.1016/j.jvir.2021.11.014. PMID 35221048

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-02): https://cdn.clinicaltrials.gov/large-docs/32/NCT07046832/Prot_SAP_000.pdf
  • Informed Consent Form (2025-05-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT07046832/ICF_001.pdf